CLINICAL TRIAL: NCT01475344
Title: A Multicenter Double-blind, Placebo Controlled, Randomized, Pilot Trial to Assess the Efficacy of Pre-hospital Administration of Fibrinogen Concentrate (FGTW) in Trauma Patients, Presumed to Bleed (FI in TIC)
Brief Title: Fibrinogen Concentrate (FGTW) in Trauma Patients, Presumed to Bleed (FI in TIC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Dietmar Fries, M.D., Coordinating and Principal Investigator, Medical University Innsbruck
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FIinTIC
Record Dates: First submitted 2011-10-27; First posted 2011-11-21 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Trauma; Massive Hemorrhage
Keywords: Trauma patient with major bleeding
MeSH Terms: conditions — Wounds and Injuries | interventions — Fibrinogen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Human Fibrinogen Concentrate (Active Comparator): Fibrinogen Concentrate will be administrated over 5 min/vial:
  Body Weight: < 30 kg / 30-60 kg / 60 - 90 kg / > 90 kg
  No. of vials: 1 vial (100 ml) / 2 vials (200 ml) / 3 vials (300 ml) / 4 vials (400 ml)
  Fibrinogen: 1.5 g / 3 g / 4.5 g / 6 g
  Immediately after admission to hospital, the patient's parameters including blood collection (see below) will be measured for the second time (T2), if applicable, after the end of administration of the study drug. Additional measurements will be made 3 hours (T3), 9 hours (T4), and 24 hours (T5), 48 hours (T6) and one week after admission (T7). 30 days after inclusion in the study, a final investigation is planned (T8).
  Interventions: Drug: Human Fibrinogen Concentrate
- Placebo (Placebo Comparator): Placebo administrated over 5 min/vial:
  Body Weight: < 30 kg / 30-60 kg / 60 - 90 kg / > 90 kg
  No. of vials: 1 vial (100 ml) / 2 vials (200 ml) / 3 vials (300 ml) / 4 vials (400 ml)
  Placebo: 1.5 g / 3 g / 4.5 g / 6 g
  Immediately after admission to hospital, the patient's parameters including blood collection (see below) will be measured for the second time (T2), if applicable, after the end of administration of the study drug. Additional measurements will be made 3 hours (T3), 9 hours (T4), and 24 hours (T5), 48 hours (T6) and one week after admission (T7). 30 days after inclusion in the study, a final investigation is planned (T8).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Human Fibrinogen Concentrate — intravenous infusion over 5 min/vial:
  Body Weight: < 30 kg / 30-60 kg / 60 - 90 kg / > 90 kg
  No. of vials: 1 vial (100 ml) / 2 vials (200 ml) / 3 vials (300 ml) / 4 vials (400 ml)
  Fibrinogen Concentrate: 1.5 g / 3 g / 4.5 g / 6 g
  Immediately after admission to hospital, the patient's parameters including blood collection (see below) will be measured for the second time (T2), if applicable, after the end of administration of the study drug. Additional measurements will be made 3 hours (T3), 9 hours (T4), and 24 hours (T5), 48 hours (T6) and one week after admission (T7). 30 days after inclusion in the study, a final investigation is planned (T8).
  Other Names: FGTW
  Arms: Human Fibrinogen Concentrate
Drug: Placebo — intravenous infusion over 5 min/vial:
  Body Weight: < 30 kg / 30-60 kg / 60 - 90 kg / > 90 kg
  No. of vials: 1 vial (100 ml) / 2 vials (200 ml) / 3 vials (300 ml) / 4 vials (400 ml)
  Placebo: 1.5 g / 3 g / 4.5 g / 6 g
  Immediately after admission to hospital, the patient's parameters including blood collection (see below) will be measured for the second time (T2), if applicable, after the end of administration of the study drug. Additional measurements will be made 3 hours (T3), 9 hours (T4), and 24 hours (T5), 48 hours (T6) and one week after admission (T7). 30 days after inclusion in the study, a final investigation is planned (T8).
  Other Names: Placebo for Fibrinogen Concentrate
  Arms: Placebo

SUMMARY:
Severe traumatized patients with visible significant bleeding and/or with clinical signs of internal significant bleeding treated by an emergency doctor of the helicopter service or the ground team will be enrolled in the study (inclusion- and exclusion criteria: see above). If a patient meets the inclusion criteria and is recruited for the study, FGTW or placebo administrated over 5 min/vial:

Body Weight: < 30 kg / 30-60 kg / 60 - 90 kg / > 90 kg

No. of vials: 1 vial (100 ml) / 2 vials (200 ml) / 3 vials (300 ml) / 4 vials (400 ml)

Fibrinogen (if applicable): 1.5 g / 3 g / 4.5 g / 6 g

DETAILED DESCRIPTION:
Severe traumatized patients with visible significant bleeding and/or with clinical signs of internal significant bleeding treated by an emergency doctor of the helicopter service or the ground team will be enrolled in the study (inclusion- and exclusion criteria: see above). If a patient meets the inclusion criteria and is recruited for the study, his baseline values on the scene (T1) will first be collected including the first blood collection as well as documentation of the clinical parameters (hemodynamics, respiratory and neurological function, etc.). Subsequently, 30 patients will be randomized to receive about 50 mg/kg BW fibrinogen concentrate (one vial for each 30 kg body weight, estimated by the emergency physician), while the other 30 patients receive placebo (also one vial including 100 ml for each 30 kg body weight). The flow rate should not exceed 100 ml within 5 minutes.

FGTW or placebo administrated over 5 min/vial:

Body Weight: < 30 kg / 30-60 kg / 60 - 90 kg / > 90 kg

No. of vials: 1 vial (100 ml) / 2 vials (200 ml) / 3 vials (300 ml) / 4 vials (400 ml)

Fibrinogen (if applicable): 1.5 g / 3 g / 4.5 g / 6 g

Immediately after admission to hospital, the patient's parameters including blood collection (see below) will be measured for the second time (T2), if applicable, after the end of administration of the study drug. Additional measurements will be made 3 hours (T3), 9 hours (T4), and 24 hours (T5), 48 hours (T6) and one week after admission (T7). 30 days after inclusion in the study, a final investigation is planned (T8).

Coagulation management after admission to hospital is depending on the specific demands of the patient and should be performed according to the recommendations of the Austrian Society for Anaesthesiology, Intensive Care Medicine and Resuscitation (ÖGARI) (http://www.oegari.at/web_files/dateiarchiv/116/key%20messages%20management%20of%20TIC%202011.pdf). Blood loss, transfusion requirements, volume therapy and coagulation therapy will be documented.

When the bleeding is under control thromboprophylaxis has to be performed according to the international standard of care earliest after 24 hours after cessation of bleeding (preferably using enoxaparin).

ELIGIBILITY:
Inclusion Criteria:

1. Trauma patient
2. Patient at the obvious age of equal or higher than 18 years of either sex
3. Major bleeding or occult bleeding with parameters of shock
4. Need for volume replacement therapy
5. Patient, who will be admitted to one of the participating hospitals

Exclusion Criteria:

1. Solely penetrating trauma
2. Solely head injury
3. In case of ongoing severe hemodynamic instability refractory to therapy (vasopressor, volume)
4. Patient with inevitable lethal course as evaluated by emergency physician
5. Need for CPR on the scene
6. Deep hypothermia (below 30°C)
7. Obviously pregnant women
8. Patient with known recent history of thromboembolic events within the last 6 months
9. Patient known to be on anticoagulant therapy
10. Patient with known refusal of a participation in this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2011-09; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change of the Fibrinogen polymerisation measured with FIBTEM® MCF | The average period for the measurement (MCF) of the primary outcome is 60 minutes . Timepoints of measurements: Emergency scene (minute 0) and arrival to the hospital (on average after 60 minutes).
  Further measurements and investigations will be done until 7 days after the hospital admission. The patient will be followed up until 30 days (final interview).

CONTACTS AND LOCATIONS:
Overall Officials: Dietmar Fries, Prof. MD, Principal Investigator — Medical University Innsbruck
Locations (16):
- Austria (11):
  - Christophorus 1, Innsbruck
  - Medical University Innsbruck, Innsbruck
  - Martin 2, Karres
  - Christophorus 14, Niederöblarn
  - AUVA Trauma Center, Salzburg
  - Christophorus 6, Salzburg
  - Alpin 2, Solden
  - NEF Telfs, Telfs
  - NAW Vöcklabruck, Vöcklabruck
  - Regional Hospital Vöcklabruck, Vöcklabruck
  - Christophorus 5, Zams
- Czechia (3):
  - Ambulace Car, Liberec
  - Krystof 18 Helicopter Base, Liberec
  - Hospital Liberec, Liberec
- Germany (2):
  - Christoph 3, Cologne
  - Cologne-Merheim Medical Center, Cologne

REFERENCES:
- [Derived] Ziegler B, Bachler M, Haberfellner H, Niederwanger C, Innerhofer P, Hell T, Kaufmann M, Maegele M, Martinowitz U, Nebl C, Oswald E, Schochl H, Schenk B, Thaler M, Treichl B, Voelckel W, Zykova I, Wimmer C, Fries D; FIinTIC study group. Efficacy of prehospital administration of fibrinogen concentrate in trauma patients bleeding or presumed to bleed (FIinTIC): A multicentre, double-blind, placebo-controlled, randomised pilot study. Eur J Anaesthesiol. 2021 Apr 1;38(4):348-357. doi: 10.1097/EJA.0000000000001366. PMID 33109923